CLINICAL TRIAL: NCT00556335
Title: A Prospective, Randomised Trial in Pneumothorax Therapy: Manual Aspiration Versus Conventional Chest Tube Drainage
Brief Title: Pneumothorax Therapy: Manual Aspiration Versus Conventional Chest Tube Drainage
Acronym: pneumothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, Dr., Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL13097.075.06
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Pneumothorax
Keywords: manual aspiration; conventional; length of stay
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- manual aspiration (Experimental): manual aspiration
  Interventions: Procedure: manual aspiration
- conventional drainage (Active Comparator): conventional drainage
  Interventions: Procedure: conventional drainage

INTERVENTIONS:
Procedure: manual aspiration — air aspiration
  Arms: manual aspiration
Procedure: conventional drainage — drainage, pneumocath
  Arms: conventional drainage

SUMMARY:
The purpose of this study is to evaluate the efficacy of manual aspiration in comparison to conventional chest tube drainage in pneumothorax therapy:

1. whether manual aspiration will shorten hospital admission.
2. whether the lung will expand by means of clinical and radiological findings.

DETAILED DESCRIPTION:
No consensus has been defined concerning the exact treatment of a first episode of SP. Literature suggests similar immediate and long-term efficacy of manual aspiration and chest tube drainage. Morbidity of manual aspiration is low and the procedure is well tolerated. Manual aspiration is safe with a complication rate of only 1 % and can be performed in the outpatient clinic in the majority of patients reducing costs. Our aim is to re - evaluate these findings with a mono-centre study with 114 patients, set-up for the first time in the Netherlands with an expectancy to confirm the former findings.

Aim of the study:

To evaluate the efficacy of manual aspiration in comparison to conventional chest tube drainage in pneumothorax therapy:

1. whether manual aspiration will shorten hospital admission.
2. whether the lung will expand by means of clinical and radiological findings.

Study design: prospective single-centre, open randomised trial.

Randomisation:

With a computer minimization program for manual aspiration or usual care with special attendance to the cause of pneumothorax (spontaneous or traumatic), the presence of smoking and gender.

Statistical analysis:

Our primary aim is to demonstrate a higher efficacy for manual aspiration in terms of a shorter admission duration (LOS) in favor of manual aspiration with similar therapy success rates. We will analyse data on an intention to treat basis. P-values below 5 % will be considered statistically significant. Normal distribution will be checked. Means (standard deviations) or medians (ranges or interquartile ranges) will be calculated and unpaired t-tests or Mann Whitney U tests will be used as appropriate to test differences in LOS. Categorical data (success rates) will be analysed using Chi2-tests. Data analysis will be performed using SPSS version 12.

Study population:

Patients with the first episode of a symptomatic pneumothorax or an asymptomatic pneumothorax with a size ≥ 20 % as estimated by Light's formula ( (1-L/H )x100 ) with an age of ≥ 18 and < 85 years.

Intervention: Manual aspiration or conventional chest tube drainage. Primary study endpoint 1. The LOS.

Secondary endpoint:

1.The success rate of each technique:

Conventional chest tube drainage; complete expansion of the lung, counteraction of the air leak and removal of the drain within 72 hours.

Manual aspiration: complete expansion and discharge within 24 hours, success rate at two weeks (continuous expansion) and one year (no recurrence of pneumothorax in the interval period after discharge between 2 weeks and 1 year).

Burden, risks and advantages associated with participation:

The risks of manual aspiration and chest tube drainage techniques are the same. Complications seem to be occur in only 1 % of the aspirations and they consist of haematothorax, retained catheter tips, subcutaneous emphysema and vasovagal reactions. The most important disadvantage is in case of an unsuccessful treatment by manual aspiration with a persisting pneumothorax. Patients in this case have to undergo the conventional tube chest drainage after all. The benefit of the investigational approach is that patients are discharged earlier from the hospital in case of success and its cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* patients with a first episode of a symptomatic pneumothorax admitted to the ER of the hospital (spontaneous or traumatic) or
* patients with an asymptomatic pneumothorax with a size of ≥ 20 % as estimated by Light's formula
* age ≥ 18 and < 85 years
* smoking is tolerated

Exclusion Criteria:

* recurrent pneumothorax
* lung fibrosis
* patients with (lung) cancer
* pregnant women
* comorbidity limiting decision making (psychiatric disease, alcohol or drug abuse)
* prior randomisation
* Marfan syndrome
* COPD patients
* tension pneumothorax
* multitrauma patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The duration of length of stay of each technique | 1 year

SECONDARY OUTCOMES:
The success rate of each technique | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: J.W. van den Berg, Dr., Study Director — Isala Klinieken department of pulmonology
Locations (1):
- Isala Klinieken, Zwolle, Netherlands

REFERENCES:
- [Background] Noppen M, Alexander P, Driesen P, Slabbynck H, Verstraeten A. Manual aspiration versus chest tube drainage in first episodes of primary spontaneous pneumothorax: a multicenter, prospective, randomized pilot study. Am J Respir Crit Care Med. 2002 May 1;165(9):1240-4. doi: 10.1164/rccm.200111-078OC. PMID 11991872
- [Derived] Parlak M, Uil SM, van den Berg JW. A prospective, randomised trial of pneumothorax therapy: manual aspiration versus conventional chest tube drainage. Respir Med. 2012 Nov;106(11):1600-5. doi: 10.1016/j.rmed.2012.08.005. Epub 2012 Aug 24. PMID 22925840